CLINICAL TRIAL: NCT00418106
Title: Early Kangaroo Holding Effects on Breast Milk Composition
Brief Title: Kangaroo Holding Effects on Breast Milk
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Amy N. Johnson, DNSc, RN, Christiana Hospital
Other Study IDs: 24211
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Premature Birth
Keywords: Premature birth; Pumping breast milk; Kangaroo holding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Mothers who are pumping breast milk and who are willing to kangaroo hold their infant.

SUMMARY:
Kangaroo holding is a skin-to-skin method of holding a baby. Many research studies have investigated the maternal and infant benefits associated with kangaroo holding. The purpose of this study is to determine if kangaroo holding a baby changes the amount and composition of breast milk pumped before and after the kangaroo holding session.

Hypotheses:

1. There is a significant difference in volume of maternal breast milk pumped after kangaroo holding premature infants as compared to maternal breast milk pumped after non-holding conditions
2. There is a significant difference in the composition of maternal breast milk pumped after kangaroo holding premature infants as compared to maternal breast milk pumped after non-holding condition.

DETAILED DESCRIPTION:
This study will address two of the overwhelming challenges in the physiologic care of premature infants in the neonatal intensive care unit (NICU) environment. The first challenge is promoting neonatal growth through providing a careful balance of nutrition to caloric expenditure for premature infants. The second challenge is supporting parents in the intensive, technology driven environment of the NICU to merge physiologic care with parental-infant interaction through touch, communication, and maternal intervention. The vast majority of mothers with premature infants express breast milk for early feedings, however milk production tends to diminish three to four weeks after delivery. The practice of skin-to-skin holding is thought to promote the mother's ability to produce breast milk, but had not been empirically tested. This study will examine the relationship of kangaroo holding on mother's breast milk production and composition.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight </= 2000 grams
* Gestational age 26-34 weeks at birth
* Medically stable at start of study
* < 14 days old at start of study

Exclusion Criteria:

* Infants receiving phototherapy
* Suspected congenital abnormalities
* Overwhelming sepsis
* Cardiac Abnormalities
* Suspected infections

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mothers of preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Breast milk production and composition | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Amy N. Johnson, DNSc, RNC, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Hospital, Newark, Delaware, United States